CLINICAL TRIAL: NCT06306040
Title: Effect of Intravenous Nalbuphine Versus Magnesium Sulfate on Emergence Agitation in Pediatric Patients Scheduled for Hypospadias Repair
Brief Title: Effect of Intravenous Nalbuphine and Magnesium Sulfate on Emergence Agitation in Pediatric
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma alzahraa Mustafa Abdelbary Thabet, Fatma Alzahraa Mustafa Abdelbary - Director, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Analgesia effect as on EA
Record Dates: First submitted 2024-02-28; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Emergence Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Intervention Model Description: * Group C (Control group n=35 ): 10 ml isotonic saline will be injected intravenously before 30 min from end of surgery
  * Group M (Magnesium sulfate group n=35 ): 30 mg/kg Magnesium sulphate diluted to 10 ml isotonic saline will be injected intravenously before 30 min from end of surgery
  * Group N (Nalbuphine group n=35 ): 0.1 mg/kg nalbuphine diluted to 10 ml isotonic saline will be injected intravenously before 30 min from end of surgery
Who Masked: Participant
Masking Description: * Group C (Control group n=35 ): 10 ml isotonic saline will be injected intravenously before 30 min from end of surgery
  * Group M (Magnesium sulfate group n=35 ): 30 mg/kg Magnesium sulphate diluted to 10 ml isotonic saline will be injected intravenously before 30 min from end of surgery
  * Group N (Nalbuphine group n=35 ): 0.1 mg/kg nalbuphine diluted to 10 ml isotonic saline will be injected intravenously before 30 min from end of surgery
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- • Group N (Nalbuphine group n=35 ) (Experimental): administrate nalbuphine 0.1 mg/kg nalbuphine diluted to 10 ml isotonic saline will be injected intravenously before 30 min from end of surgery (injected once) dose
  Interventions: Drug: Nalbuphine Versus Magnesium Sulfate
- • Group M (Magnesium sulfate group n=35 ) (Experimental): administrate magnesium sulfate once 30 mg/kg Magnesium sulphate diluted to 10 ml isotonic saline will be injected intravenously before 30 min from end of surgery
  Interventions: Drug: Nalbuphine Versus Magnesium Sulfate
- Group C (Control group n=35 ): (Experimental): administrate 10 ml isotonic saline will be injected intravenously before 30 min from end of surgery
  Interventions: Drug: Nalbuphine Versus Magnesium Sulfate

INTERVENTIONS:
Drug: Nalbuphine Versus Magnesium Sulfate — Nalbuphine is a synthetic opioid receptor agonist-antagonist (agonist К receptor, antagonistic part μ receptor) that can produce a central analgesic effect and partial sedation. Nalbuphine is a medication that is indicated for moderate to severe pain where the patient requires an opioid agent, and other alternative treatments have been insufficient. The inhibitory effect of nalbuphine on respiration is slight and it has a capping effect. Owing to these advantages, it is widely used in pediatric surgical analgesia.
  Magnesium sulphate, an antagonist of N-methyl-D-aspartate (NMDA) glutamate receptors, has been reported to improve hypo-magnesia and pre-eclampsia. Recently, magnesium sulphate has been gradually used as an adjuvant for sedation and analgesia during general anesthesia. Magnesium sulphate is a medication used to manage and treat multiple clinical conditions.
  Other Names: analgesic effect on emergency agitation

SUMMARY:
• Primary outcome: Measure The incidence of EA in children undergoing to hypospadias repair under general anesthesia is considered using Pediatric Anesthesia Emergence Delirium (PAED) scales.

• Secondary outcome:

* Therefore, we designed a prospective, randomized, double-blind, single center study to investigate whether nalbuphine and/or magnesium sulphate can prevent EA after hypospadias repair in children under general anesthesia. In addition, the characteristics of anesthesia recovery and the incidence of adverse effects will also be evaluated in this study. Post-operative extubating time, interaction time, open eye time and emergence time. incidence of post-operative vomiting (PONV), laryngospasm, breath-holding, coughing, oxygen desaturation, and cardiac arrhythmias.
* Face, Legs, Activity, Cry and Consola Bility (FLACC) scale is used to determine post-operative pain score
* Parental satisfaction scores

DETAILED DESCRIPTION:
Emergence agitation (EA), also referred to as emergence delirium, emergence excitement or inadequate emergence, is a frequent post-operative complication in pediatric patients receiving inhalational anesthetics. It's defined as an acute and fluctuating alteration of mental state and manifesting as agitation, confusion, disorientation, and hyperactivity during the transition from unconsciousness to full wakefulness. The incidence of EA is reported to be up to 20% in adult patients and up to 80% in children.

Although EA is self-limiting, it can induce potential problems in children, such as self-injury, bleeding and cracking of the wound, falling off of the indwelling catheter, and falling off of the bed, which can cause some difficulties for medical staff and serious anxiety for family members. In addition, children with EA are at a higher risk of post-hospitalization behavioral changes, which may last longer. Furthermore, EA treatment increases the burden on healthcare providers and increases the medical expenses of patients. EA commonly occurs after the most common surgeries in children like adenoidectomy, tonsillectomy, hernioplasty and hypospadias repair. Therefore, implementing effective measures to prevent EA in children undergoing these types of surgeries is crucial. Although the underlying mechanisms of EA remain unclear, the mechanisms may be related to pre-operative anxiety, inhaled anesthetics (sevoflurane or desflurane), surgery type (ophthalmology or otolaryngology procedure), and younger age.

Some pharmacological interventions have been used to prevent and treat EA. Previous studies have demonstrated that propofol, benzodiazepines, α2 agonists, and opioids can prevent EA in children to varying degrees. However, these medications may lead to respiratory depression, delay in anesthesia recovery and post-anesthesia care unit stay, and other adverse reactions. Thus, the most favorable prophylactic treatment to decrease such an incidence remains unknown, and the ideal approaches to prevent EA merit further exploration.

Nalbuphine is a synthetic opioid receptor agonist-antagonist (agonist К receptor, antagonistic part μ receptor) that can produce a central analgesic effect and partial sedation. Nalbuphine is a medication that is indicated for moderate to severe pain where the patient requires an opioid agent, and other alternative treatments have been insufficient. The inhibitory effect of nalbuphine on respiration is slight and it has a capping effect. Owing to these advantages, it is widely used in pediatric surgical analgesia.

Magnesium sulphate, an antagonist of N-methyl-D-aspartate (NMDA) glutamate receptors, has been reported to improve hypo-magnesia and pre-eclampsia. Recently, magnesium sulphate has been gradually used as an adjuvant for sedation and analgesia during general anesthesia. Magnesium sulphate is a medication used to manage and treat multiple clinical conditions.

ELIGIBILITY:
Inclusion Criteria:

* • Weight: 10 - 38 kg.

  * Age: 3-7 years.
  * ASA physical status: I-II.
  * Operation: elective hypospadias repair under general anesthesia

Exclusion Criteria:

* • Parent's refusal.

  * Anticipated difficult airway.
  * Active respiratory illness (cough, fever, rhinorrhea) on the day of anesthesia.
  * History of developmental delay or mental retardation or any neurological disease.
  * Known hypersensitivity to any drug used in this study.
  * Children with co-morbid conditions like congenital heart disease, respiratory pathology, central nervous system disorders or renal pathology

Ages: 3 Years to 7 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — name of patient gender exposure on surgery only male participants are being due to surgery is hypospadias repair.
Enrollment: 105 (Estimated)
Dates: Start 2024-04-02 (Estimated); Primary Completion 2024-11-03 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
compare between analgesia effect on pediatric patient | baseline
  Measure The incidence of EA in children undergoing to hypospadias repair under general anesthesia is considered using Pediatric Anesthesia Emergence Delirium (PAED) scales.

CONTACTS AND LOCATIONS:
Overall Officials: Abualauon M Mohamed Abdelmohsen Rashwan, Lecturer, Study Director — Assiut University

REFERENCES:
- [Background] Lee SJ, Sung TY. Emergence agitation: current knowledge and unresolved questions. Korean J Anesthesiol. 2020 Dec;73(6):471-485. doi: 10.4097/kja.20097. Epub 2020 Mar 25. PMID 32209961
- [Background] Dahmani S, Stany I, Brasher C, Lejeune C, Bruneau B, Wood C, Nivoche Y, Constant I, Murat I. Pharmacological prevention of sevoflurane- and desflurane-related emergence agitation in children: a meta-analysis of published studies. Br J Anaesth. 2010 Feb;104(2):216-23. doi: 10.1093/bja/aep376. Epub 2010 Jan 3. PMID 20047899
- [Background] Yu D, Chai W, Sun X, Yao L. Emergence agitation in adults: risk factors in 2,000 patients. Can J Anaesth. 2010 Sep;57(9):843-8. doi: 10.1007/s12630-010-9338-9. Epub 2010 Jun 5. PMID 20526708
- [Background] Choi EK, Park S, Park KB, Kwak KH, Park S. Postoperative emergence agitation and intraoperative sevoflurane sedation under caudal block in children: a randomized comparison of two sevoflurane doses. Anesth Pain Med (Seoul). 2019 Oct 31;14(4):434-440. doi: 10.17085/apm.2019.14.4.434. PMID 33329774
- [Background] Zhang YZ, Wei XL, Tang B, Qin YY, Ou M, Jiang XH, Tan YF, Ye MY. The Effects of Different Doses of Alfentanil and Dexmedetomidine on Prevention of Emergence Agitation in Pediatric Tonsillectomy and Adenoidectomy Surgery. Front Pharmacol. 2022 Feb 2;13:648802. doi: 10.3389/fphar.2022.648802. eCollection 2022. PMID 35185554
- [Background] Kim J, Byun SH, Kim JW, Kim JY, Kim YJ, Choi N, Lee BS, Yu S, Kim E. Behavioral changes after hospital discharge in preschool children experiencing emergence delirium after general anesthesia: A prospective observational study. Paediatr Anaesth. 2021 Oct;31(10):1056-1064. doi: 10.1111/pan.14259. Epub 2021 Aug 6. PMID 34309126
- [Background] Voepel-Lewis T, Malviya S, Tait AR. A prospective cohort study of emergence agitation in the pediatric postanesthesia care unit. Anesth Analg. 2003 Jun;96(6):1625-1630. doi: 10.1213/01.ANE.0000062522.21048.61. PMID 12760985
- [Background] Mason KP. Paediatric emergence delirium: a comprehensive review and interpretation of the literature. Br J Anaesth. 2017 Mar 1;118(3):335-343. doi: 10.1093/bja/aew477. PMID 28203739
- [Background] Kanaya A. Emergence agitation in children: risk factors, prevention, and treatment. J Anesth. 2016 Apr;30(2):261-7. doi: 10.1007/s00540-015-2098-5. Epub 2015 Nov 24. PMID 26601849
- [Background] Jalili S, Esmaeeili A, Kamali K, Rashtchi V. Comparison of effects of propofol and ketofol (Ketamine-Propofol mixture) on emergence agitation in children undergoing tonsillectomy. Afr Health Sci. 2019 Mar;19(1):1736-1744. doi: 10.4314/ahs.v19i1.50. PMID 31149004
- [Background] Kawai M, Kurata S, Sanuki T, Mishima G, Kiriishi K, Watanabe T, Ozaki-Honda Y, Yoshida M, Okayasu I, Ayuse T, Tanoue N, Ayuse T. The effect of midazolam administration for the prevention of emergence agitation in pediatric patients with extreme fear and non-cooperation undergoing dental treatment under sevoflurane anesthesia, a double-blind, randomized study. Drug Des Devel Ther. 2019 May 17;13:1729-1737. doi: 10.2147/DDDT.S198123. eCollection 2019. PMID 31190751
- [Background] Kim SY, Kim JM, Lee JH, Song BM, Koo BN. Efficacy of intraoperative dexmedetomidine infusion on emergence agitation and quality of recovery after nasal surgery. Br J Anaesth. 2013 Aug;111(2):222-8. doi: 10.1093/bja/aet056. Epub 2013 Mar 22. PMID 23524149
- [Background] Cravero JP, Beach M, Thyr B, Whalen K. The effect of small dose fentanyl on the emergence characteristics of pediatric patients after sevoflurane anesthesia without surgery. Anesth Analg. 2003 Aug;97(2):364-367. doi: 10.1213/01.ANE.0000070227.78670.43. PMID 12873918
- [Background] Kubica-Cielinska A, Zielinska M. The use of nalbuphine in paediatric anaesthesia. Anaesthesiol Intensive Ther. 2015;47(3):252-6. doi: 10.5603/AIT.2015.0036. PMID 26165241
- [Background] Shin D, Kim S, Kim CS, Kim HS. Postoperative pain management using intravenous patient-controlled analgesia for pediatric patients. J Craniofac Surg. 2001 Mar;12(2):129-33. doi: 10.1097/00001665-200103000-00007. PMID 11314621
- [Background] Urits I, Jung JW, Amgalan A, Fortier L, Anya A, Wesp B, Orhurhu V, Cornett EM, Kaye AD, Imani F, Varrassi G, Liu H, Viswanath O. Utilization of Magnesium for the Treatment of Chronic Pain. Anesth Pain Med. 2021 Feb 6;11(1):e112348. doi: 10.5812/aapm.112348. eCollection 2021 Feb. PMID 34221945
- [Background] Sullivan M, Cunningham K, Angras K, Mackeen AD. Duration of postpartum magnesium sulfate for seizure prophylaxis in women with preeclampsia: a systematic review and meta-analysis. J Matern Fetal Neonatal Med. 2022 Dec;35(25):7188-7193. doi: 10.1080/14767058.2021.1946505. Epub 2021 Jun 30. PMID 34187284
- [Background] Lysakowski C, Dumont L, Czarnetzki C, Tramer MR. Magnesium as an adjuvant to postoperative analgesia: a systematic review of randomized trials. Anesth Analg. 2007 Jun;104(6):1532-9, table of contents. doi: 10.1213/01.ane.0000261250.59984.cd. PMID 17513654
- [Background] Abdulatif M, Ahmed A, Mukhtar A, Badawy S. The effect of magnesium sulphate infusion on the incidence and severity of emergence agitation in children undergoing adenotonsillectomy using sevoflurane anaesthesia. Anaesthesia. 2013 Oct;68(10):1045-52. doi: 10.1111/anae.12380. Epub 2013 Aug 3. PMID 23909742
- [Background] Xie M, Li XK, Peng Y. Magnesium sulfate for postoperative complications in children undergoing tonsillectomies: a systematic review and meta-analysis. J Evid Based Med. 2017 Feb;10(1):16-25. doi: 10.1111/jebm.12230. PMID 27787936
- [Background] Albrecht E, Kirkham KR, Liu SS, Brull R. Peri-operative intravenous administration of magnesium sulphate and postoperative pain: a meta-analysis. Anaesthesia. 2013 Jan;68(1):79-90. doi: 10.1111/j.1365-2044.2012.07335.x. Epub 2012 Nov 1. PMID 23121612
- [Background] Sikich N, Lerman J. Development and psychometric evaluation of the pediatric anesthesia emergence delirium scale. Anesthesiology. 2004 May;100(5):1138-45. doi: 10.1097/00000542-200405000-00015. PMID 15114210
- [Background] Malviya S, Voepel-Lewis T, Burke C, Merkel S, Tait AR. The revised FLACC observational pain tool: improved reliability and validity for pain assessment in children with cognitive impairment. Paediatr Anaesth. 2006 Mar;16(3):258-65. doi: 10.1111/j.1460-9592.2005.01773.x. PMID 16490089
- [Background] White PF, Song D. New criteria for fast-tracking after outpatient anesthesia: a comparison with the modified Aldrete's scoring system. Anesth Analg. 1999 May;88(5):1069-72. doi: 10.1097/00000539-199905000-00018. No abstract available. PMID 10320170